CLINICAL TRIAL: NCT06936878
Title: BOLSTER: Strengthening Patient and Caregiver Supports in Advanced Gynecologic and Gastrointestinal Cancers
Brief Title: BOLSTER: Learning New Skills to Thrive
Acronym: BOLSTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-523; R01CA270040-01A1 (NIH)
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Cancer; Gynecologic Cancer; Advanced Cancer
Keywords: Gastrointestinal Cancer; Gynecologic Cancer; Advanced Cancer; Advanced Gastrointestinal Cancer; Advanced Gynecologic Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Usual Care (No Intervention): Participants and their care partners (a family member or loved one involved in their care) will be randomized in a 1:1 fashion and stratified by institution and cancer type and will complete:
  * Baseline visit
  * Standard-of-care oncology appointments
  * Access to nurse and specialist appointments
  * 6 week survey
  * 12 week survey
- Arm 2: Bolster Program (Experimental): Patients and their care partners (a family member or loved one involved in their care) will be randomized in a 1:1 fashion and stratified by institution and cancer type and will complete:
  * Baseline visit
  * 6 telehealth sessions with a nurse for patients and their care partners
  * 2 brief telehealth sessions for care partners.
  * Access to the Bolster Program website with tailored educational materials
  * 6 week survey
  * 12 week survey
  Interventions: Behavioral: BOLSTER Program

INTERVENTIONS:
Behavioral: BOLSTER Program — This supportive care program includes six telehealth sessions led by a trained nurse to help patients with advanced gynecological or gastrointestinal cancers and their care partners build skills, manage symptoms, and cope with challenges. Two additional sessions will be help support care partners. Participants will also get access to the BOLSTER website, which offers personalized educational materials to support their well-being
  Other Names: BOLSTER
  Arms: Arm 2: Bolster Program

SUMMARY:
This research study is evaluating a new program called Building Out Lifelines for Safety, Trust, Empowerment, and Renewal or (BOLSTER), which was designed to support participants with a gynecological or gastrointestinal cancer and new and complex care needs.

DETAILED DESCRIPTION:
This multi-center, randomized trial is to test the efficacy of the BOLSTER Program and to improve participant quality of life (QOL), alleviate symptoms, reduce burden, and decrease the need for hospital care in participants with complex care needs from advanced gastrointestinal and gynecologic (GI/GYN) cancers.

The research study procedures include screening for eligibility, questionnaires, and telehealth visits.

Participation in this research study is expected to last about 12 weeks.

About 300 dyads (patients with family caregivers) are expected to participate in this research study.

The National Cancer Institute is funding this research study by providing funding.

ELIGIBILITY:
Participant Inclusion Criteria:

* Age ≥18 years
* Currently hospitalized with skilled care need or have acquired a new skilled care need as an outpatient
* Diagnosed with advanced gastrointestinal cancer (esophageal, gastric, pancreatic, hepatobiliary, colorectal, unknown GI primary, anal) or advanced gynecologic cancer (ovarian, endometrial, cervical, vaginal, vulvar)
* Has a complex care need (e.g., ostomy, ileostomy, urostomy, nephrostomy, biliary drain, venting gastric tube, feeding tube, intraabdominal or pleural catheter, wound VAC)
* Plans to receive ongoing cancer treatment
* Has a family caregiver or friend (hereafter designated family caregiver) willing to participate
* Able to speak and read English or Spanish (self-report)
* Are willing to be audio-recorded
* Have the cognitive/physical ability to participate in a 60-minute interview

Family or Caregiver Inclusion Criteria:

* Age ≥ 18 years
* Identified by a patient (as defined above) as a family or friend who is involved in their care.
* Willing to participate in study visits
* Willing to be audio recorded

Participant Exclusion Criteria:

* Has cognitive impairments (as determined by the patient's oncologist)
* Planning to enroll in hospice
* Unable to complete baseline survey
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Family or Caregiver Exclusion Criteria:

* Unable to complete baseline survey
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the FACT-G, a 27-item scale designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 108. Higher scores indicate better quality of life.
Change in FACT-G Score From Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the FACT-G, a 27-item scale designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 108. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Change in FACT-G Score From Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the FACT-G, a 27-item scale designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 108. Higher scores indicate better quality of life.
Change in FACT-G Score From Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the FACT-G, a 27-item scale designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 108. Higher scores indicate better quality of life.
Change in Functional Assessment of Cancer Therapy-General 7 item Version (FACT-G7) Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the FACT-G7, a 7-item designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer in the past 7 days. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 28. A higher score indicates better quality of life.
Change in FACT-G7 Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the FACT-G7, a 7-item designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer in the past 7 days. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 28. A higher score indicates better quality of life.
Change in FACT-G7 Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the FACT-G7, a 7-item designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer in the past 7 days. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 28. A higher score indicates better quality of life.
Change in FACT-G7 Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the FACT-G7, a 7-item designed to measure physical, emotional, social, functional, and family well-being in patients with life-limiting cancer in the past 7 days. Answers are rated on a 5-point Likert scale from 0 "Not At All" to 4 "Very Much" with a total scores range of 0 to 28. A higher score indicates better quality of life.
Change in Participant Self-Efficacy for Managing Chronic Conditions Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the Self-Efficacy for Managing Chronic Conditions - Short Form 4a, an 8-item measure for determining managements of symptoms and medications. Answers are rated on a 5-point Likert scale from 1 "I am not at all confident" to 5 "I am very confident" with a total scores range of 0 to 40. A higher score indicates greater self-efficacy.
Change in Participant Self-Efficacy for Managing Chronic Conditions Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the Self-Efficacy for Managing Chronic Conditions - Short Form 4a, an 8-item measure for determining managements of symptoms and medications. Answers are rated on a 5-point Likert scale from 1 "I am not at all confident" to 5 "I am very confident" with a total scores range of 0 to 40. A higher score indicates greater self-efficacy.
Change in Participant Self-Efficacy for Managing Chronic Conditions Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Care Needs and Managing Medications and Treatment. The Managing Care Needs (7 items) and Managing Medications and Treatment - Short Form 4a (6 items) evaluate confidence in handling medical care, including managing devices, medications, and symptoms. Responses are rated on a 5-point Likert scale from 1 ("Not at all confident") to 5 ("Very confident"), with higher scores indicating greater self-efficacy.
Change in Participant Self-Efficacy for Managing Chronic Conditions Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Care Needs and Managing Medications and Treatment. The Managing Care Needs (7 items) and Managing Medications and Treatment - Short Form 4a (6 items) evaluate confidence in handling medical care, including managing devices, medications, and symptoms. Responses are rated on a 5-point Likert scale from 1 ("Not at all confident") to 5 ("Very confident"), with higher scores indicating greater self-efficacy.
Change in Health Care Utilization from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Defined as the numeric value of the frequency of health care utilization by participant and collected by the Health Care Utilization Report, which is a log that covers the previous 12 weeks and collects emergency room visits, hospitalizations, and rehabilitation admissions.
Change in Health Care Utilization from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Defined as the numeric value of the frequency of health care utilization by participant and collected by the Health Care Utilization Report, which is a log that covers the previous 12 weeks and collects emergency room visits, hospitalizations, and rehabilitation admissions.
Change in Advanced care planning (ACP) from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  ACP measures a patient's preferences, understanding, and preparedness for future medical care, as documented in the electronic health record.
Change in Advanced care planning (ACP) from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  ACP measures a patient's preferences, understanding, and preparedness for future medical care, as documented in the electronic health record.
Change in Participant Hospital Anxiety and Depression (HADS) Anxiety Subscale Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Participant HADS Anxiety Subscale Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Participant HADS Anxiety Subscale Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Participant HADS Anxiety Subscale Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Participant HADS Depression Subscale Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Participant HADS Depression Subscale Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Participant HADS Depression Subscale Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Participant HADS Depression Subscale Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Caregiver Perception of Quality of End-of-Life Care | Up to 12 weeks
  Caregiver perception of end-of-life care will be assessed through a validated after-death bereaved family interview, evaluating healthcare utilization, quality of care, symptom management, and goal attainment.
Change in Caregiver Short Form ZARIT Burden Interview (ZBI-12) Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the Short Form ZARIT Burden Interview, a 12-item measure rated on a 5-point Likert scale with answers ranging from 0 "Never" to 4 "Nearly always." A total scores range is 0 to 48 with a higher score indicating higher caregiver burden.
Change in Caregiver ZBI-12 Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the Short Form ZARIT Burden Interview, a 12-item measure rated on a 5-point Likert scale with answers ranging from 0 "Never" to 4 "Nearly always." A total scores range is 0 to 48 with a higher score indicating higher caregiver burden.
Change in Caregiver ZBI-12 Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the Short Form ZARIT Burden Interview, a 12-item measure rated on a 5-point Likert scale with answers ranging from 0 "Never" to 4 "Nearly always." A total scores range is 0 to 48 with a higher score indicating higher caregiver burden.
Change in Caregiver ZBI-12 Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the Short Form ZARIT Burden Interview, a 12-item measure rated on a 5-point Likert scale with answers ranging from 0 "Never" to 4 "Nearly always." A total scores range is 0 to 48 with a higher score indicating higher caregiver burden.
Change in Caregiver HADS Anxiety Subscale Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Caregiver HADS Anxiety Subscale Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Caregiver HADS Anxiety Subscale Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Caregiver HADS Anxiety Subscale Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the Anxiety Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for anxiety.
Change in Caregiver HADS Depression Subscale Score from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Caregiver HADS Depression Subscale Score from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Caregiver HADS Depression Subscale Score from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Caregiver HADS Depression Subscale Score from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  Assessed by the Depression Subscale of the HADS questionnaire, a 7-item survey with answers scored on a 0-3 point scale. A total scores range is 0 - 21 with a higher score indicating increasing abnormality (or caseness) for depression.
Change in Caregiver-Patient Activation from Baseline to Week 6 (Arm 1) | Baseline to 6 weeks post-discharge
  The Caregiver Patient Activation Survey is a 10-item survey used to measure a caregiver's knowledge, skills, confidence, and willingness to advocate for and support a patient's healthcare needs. It assesses the caregiver's ability to navigate the healthcare system, communicate with providers, manage medications, and ensure adherence to treatment plans.
Change in Caregiver-Patient Activation from Baseline to Week 6 (Arm 2) | Baseline to 6 weeks post-discharge
  The Caregiver Patient Activation Survey is a 10-item survey used to measure a caregiver's knowledge, skills, confidence, and willingness to advocate for and support a patient's healthcare needs. It assesses the caregiver's ability to navigate the healthcare system, communicate with providers, manage medications, and ensure adherence to treatment plans.
Change in Caregiver-Patient Activation from Baseline to Week 12 (Arm 1) | Baseline to 12 weeks post-discharge
  The Caregiver Patient Activation Survey is a 10-item survey used to measure a caregiver's knowledge, skills, confidence, and willingness to advocate for and support a patient's healthcare needs. It assesses the caregiver's ability to navigate the healthcare system, communicate with providers, manage medications, and ensure adherence to treatment plans.
Change in Caregiver-Patient Activation from Baseline to Week 12 (Arm 2) | Baseline to 12 weeks post-discharge
  The Caregiver Patient Activation Survey is a 10-item survey used to measure a caregiver's knowledge, skills, confidence, and willingness to advocate for and support a patient's healthcare needs. It assesses the caregiver's ability to navigate the healthcare system, communicate with providers, manage medications, and ensure adherence to treatment plans.

CONTACTS AND LOCATIONS:
Overall Officials: Alexi Wright, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu